CLINICAL TRIAL: NCT06783088
Title: Quantification With Lutetium-177 on Cadmium-Zinc-Telluride Camera 3D
Acronym: QUADO
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, IMBERT Laetitia, Principal investigator, Central Hospital, Nancy, France
Other Study IDs: 2024PI251
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main of this study is to demonstrate the feasibility of carrying out quantitative acquisitions regardless of the energy peak considered (113 keV (kiloelectronVolts) or 208 keV or a combination of the 2 energy peaks). A study on phantom will optimise the reconstruction parameters. These parameters will then be applied to a population of patients who have already benefited from a recording on a 3D CZT camera (retrospective data).

DETAILED DESCRIPTION:
Lutetium 177 is a beta emitter - and is used in therapy. It also emits during its radioactive decay, two gamma photons of energy 113 and 208 keV allowing to produce images. The dosimetry committee of the European Association for Nuclear Medicine (EANM) recommends using only the peak at 208 keV to obtain so-called quantitative images using a conventional camera also called an Anger camera.

For several years, new semiconductor cameras (CZT cameras) have been available in nuclear medicine departments. They offer better performances particularly in terms of detection sensitivity and energy resolution. The nuclear medicine team has already carried out studies with Lutetium-177 with these semiconductor cameras on phantoms as well as dosimetry studies after treatment using Lutetium-177.

This study should demonstrate the feasibility of carrying out quantitative acquisitions regardless of the energy peak considered (113 keV or 208 keV or a combination of the 2 energy peaks). A study on phantom will optimise the reconstruction parameters. These parameters will then be applied to a population of patients who have already benefited from a recording on a 3D CZT camera (Retrospective data).

ELIGIBILITY:
It is a retrospective study and the criteria to collect the imaging are:

Inclusion Criteria:

Patients treated by at least one cure of lutetium vipivotide tetraxetan with imaging

Exclusion Criteria:

Patient having sent an objection to the use of their data

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have already benefited from at least one course of lutetium vipivotide tetraxetan and a recording on a 3D Cadmium Zinc Telluride camera made the day after treatment (image on Day N°1, Day 0 being the day of treatment administration)
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Demonstrate that the quantification of images obtained with the 113 keV peak is equivalent to the quantification obtained with the 208 keV peak. | one day
  Measurement of contrast coefficients and metabolic volumes on reconstructed images

CONTACTS AND LOCATIONS:
Locations (1):
- Chru Nancy, Vandœuvre-lès-Nancy, France